CLINICAL TRIAL: NCT06625320
Title: RASolute 302: A Phase 3 Multicenter, Open-label, Randomized Study of Daraxonrasib (RMC-6236) Versus Investigator's Choice of Standard of Care Therapy in Patients With Previously Treated Metastatic Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Phase 3 Study of Daraxonrasib (RMC-6236) in Patients With Previously Treated Metastatic Pancreatic Ductal Adenocarcinoma (PDAC)
Acronym: RASolute 302
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6236-302
Record Dates: First submitted 2024-09-20; First posted 2024-10-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; PDAC; PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer; PDAC; Pancreatic Ductal Adenocarcinoma; RAS; KRAS; NRAS; HRAS; RAS Wild-Type; RAS Q61 Mutation; RAS G12 Mutation; RAS G13 Mutation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Irinotecan; irinotecan sucrosofate; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RMC-6236 (Experimental): Study drug
  Interventions: Drug: RMC-6236
- Investigator's choice of standard of care therapy (Active Comparator): Patients randomized to Investigator's choice of standard of care chemotherapy will receive one of the following four treatments:
  * Gemcitabine and nab-paclitaxel (GnP)
  * Oxaliplatin, leucovorin, irinotecan, and 5-FU (Modified FOLFIRINOX: mFOLFIRINOX)
  * Liposomal irinotecan (Nal-IRI + 5-FU/LV)
  * Oxaliplatin, leucovorin and 5-FU IV (FOLFOX)
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: Irinotecan; Drug: Liposomal irinotecan; Drug: 5-fluorouracil; Drug: leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: RMC-6236 — Oral Tablets
  Arms: RMC-6236
Drug: Gemcitabine — intravenous (IV) infusion
  Arms: Investigator's choice of standard of care therapy
Drug: nab-paclitaxel — IV infusion
  Arms: Investigator's choice of standard of care therapy
Drug: Irinotecan — IV infusion
  Arms: Investigator's choice of standard of care therapy
Drug: Liposomal irinotecan — IV infusion
  Arms: Investigator's choice of standard of care therapy
Drug: 5-fluorouracil — IV infusion
  Arms: Investigator's choice of standard of care therapy
Drug: leucovorin — IV infusion
  Arms: Investigator's choice of standard of care therapy
Drug: Oxaliplatin — IV infusion
  Arms: Investigator's choice of standard of care therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a novel RAS(ON) inhibitor compared to standard(s) of care (SOC) treatment.

DETAILED DESCRIPTION:
This is a global, randomized, open-label, Phase 3 study designed to evaluate whether treatment with RMC-6236 will improve progression free survival (PFS) or overall survival (OS) compared to Investigator's choice of standard of care chemotherapy in patients with metastatic PDAC who were previously treated with one prior line of therapy with 5-fluorouracil (5-FU) based or gemcitabine-based regimen.

Patients will be randomized in a 1:1 ratio to receive RMC-6236 (Arm A) or Investigator's choice of standard of care chemotherapy (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and has provided informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Histologically or cytologically confirmed PDAC with metastatic disease.
* Measurable disease per RECIST 1.1.
* Adequate organ function (bone marrow, liver, kidney, coagulation)
* Documented RAS mutation status, either mutant or wild-type. RAS mutations defined as nonsynonymous mutations in KRAS, NRAS, or HRAS at codons 12, 13, or 61 (G12, G13, or Q61).
* Able to take oral medications.

Exclusion Criteria:

* Prior therapy with direct RAS-targeted therapy (eg. degraders and/or inhibitors).
* History of or known central nervous system metastatic disease.
* Any conditions that may affect the ability to take or absorb study treatment
* Major surgery within 4 weeks prior to randomization.
* Patient is unable or unwilling to comply with protocol-required study visits or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in the RAS G12-mutant population | Up to approximately 3 years
  PFS is defined as the time from randomization until disease progression or death from any cause, whichever occurs first. Progression is per response evaluation criteria in solid tumors (RECIST) v1.1 and as assessed by blinded independent central review (BICR)
Overall survival (OS) in the RAS G12-mutant population | Up to approximately 3 years
  OS is defined as the time from randomization until death from any cause.

SECONDARY OUTCOMES:
PFS in the all-patient population | Up to approximately 3 years
  PFS is defined as the time from randomization until disease progression or death from any cause, whichever occurs first. Progression is per RECIST v1.1 and as assessed by BICR.
OS in the all-patient population | Up to approximately 3 years
  OS is defined as the time from randomization until death from any cause.
Objective response in the RAS G12 and all-patient populations | Up to approximately 3 years
  Objective response is defined as partial response (PR) or completed response (CR) per RECIST v1.1, assessed by BICR.
Time to deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Pancreatic Cancer Module (EORTC QLQ-PAN26) in the RAS G12 and all-patient populations | Up to approximately 3 years
  TTD is defined as the time from randomization to the first occurrence of deterioration as defined by a change of at least 10 points, or death, whichever occurs first, in each subscale in EORTC QLQ-PAN26.
Time to deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in the RAS G12 and all-patient populations | Up to approximately 3 years
  TTD is defined as the time from randomization to the first occurrence of deterioration as defined by a change of at least 10 points, or death, whichever occurs first, in each subscale and global QoL score in EORTC QLQ-C30.
Objective response per investigator in RAS G12 and all- patient populations | Up to approximately 3 years
  Objective response is defined as PR or CR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by the investigator.
Duration of response (DOR) in RAS G12 and all-patient populations | Up to approximately 3 years
  DOR is defined as time from first evidence of objective response (PR or CR) to disease progression or death due to any cause, whichever occurs first, as assessed by BICR and by the investigator.
Time to response (TTR) in RAS G12 and all-patient populations | Up to approximately 3 years
  TTR is defined as time from randomization to first evidence of objective response (PR or CR), as assessed by BICR and by the investigator.
Percentage of patients with adverse events (AEs) | Up to approximately 3 years
Pharmacokinetics of RMC-6236 in RAS G12 and all-patient populations | Up to approximately 3 years
  Pharmacokinetics are defined by blood concentrations of RMC-6236 over time.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Revolution Medicines
Locations (60):
- United States (37):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Cancer Center - Phoenix, Phoenix, Arizona
  - City of Hope-Duarte, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - UC San Diego Health Moores Cancer Center, San Diego, California
  - Mission Hall UCSF, San Francisco, California
  - Rocky Mountain Cancer, Aurora, Colorado
  - Mayo Clinic Cancer Center - Florida, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Cancer Care Centers of Brevard Inc, Palm Bay, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - The University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Lagone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Abramson Cancer Center Clinical Research Unit, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute (Tennessee), Nashville, Tennessee
  - Texas Oncology Sammons, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Central South, Irving, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Centre Eugene Marquis, Rennes
  - Hopital Paul Brousse, Villejuif
  - Gustave Roussy, Villejuif
- Germany (4):
  - Charité Universitätsmedizin, Campus Berlin Mitte, Berlin
  - Nationales Centrum fur, Heidelberg
  - Universitatsklinikum Ulm, Zentru, München
  - Universitatsklinikum Ulm, Ulm
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO-Istituto Europeo di Oncologia, Milan
  - IOV-Istituto Oncologico, Padua
  - Azienda Ospedaliera, Pisa
- Japan (6):
  - National Cancer Center, Chiba
  - Aichi Cancer Center, Nagoya
  - Osaka International Cancer, Osaka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Pan-American Center for Oncology Trials, San Juan, Puerto Rico
- Spain (4):
  - Hospital Unversitari, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico de Valencia, Valencia